CLINICAL TRIAL: NCT07143721
Title: Comparison of the Effect of Different Inspiratory Loads on Diaphragmatic Function in Healthy Individuals
Status: Active, not recruiting | Type: Observational
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Eva María Lantarón Caeiro, principal investigator, University of Vigo
Other Study IDs: Muscle training
Record Dates: First submitted 2025-06-24; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: Diaphragm ultrasound; inspiratory muscle training; respiratory biomechanics; muscle mobility; lung function; breathing exercise; respiratory evaluation; muscle thickness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy adults undergoing inspiratory muscle training at varying intensities: Ultrasound assessment of diaphragm movement and thickness, spirometry, maximum inspiratory pressure measurement, breathing exercises at different load intensities.

SUMMARY:
This pilot study aims to evaluate how the diaphragm responds to different inspiratory muscle training loads using ultrasound in healthy individuals. The observational, cross-sectional research seeks to determine whether ultrasound measurements of diaphragm movement and thickness can more effectively guide load prescription, thereby optimizing the benefits of inspiratory training. Twenty healthy participants, of both sexes, aged 18 to 35 years, will be recruited through outreach at the Faculty of Physiotherapy at the University of Vigo. The assessment will include spirometry, maximum inspiratory pressure (MIP) measurement, and ultrasound evaluations of the diaphragm at various loads (10%, 30%, 50%, and 70% of the MIP). Data will be analyzed to understand how diaphragm mobility, thickness, and contraction velocity vary according to load, with the goal of improving training prescription and adjustment. The study adheres to the ethical principles of the Declaration of Helsinki and ensures strict confidentiality and participant anonymity. The results will contribute to the understanding of non-invasive diaphragm assessment and its role in enhancing respiratory and physical performance.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults aged 18 to 35 years

No history of neuromuscular, cardiovascular, respiratory, or musculoskeletal diseases that could limit participation

Not currently on medication affecting muscle function

Willing to provide informed consent

Exclusion Criteria:

Pregnant women

Recent thoracic or abdominal trauma (within the last 3 months)

Respiratory symptoms in the last two weeks

Conditions preventing performing forced inspiratory maneuvers

Recent respiratory muscle training (within the last 6 months)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers aged 18-35 years, without any history of respiratory or musculoskeletal diseases, and without conditions that could affect diaphragmatic function assessment.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in diaphragmatic excursion during inspiratory muscle training at varying loads | Day 2: Baseline; Immediately after 10% MIP; Immediately after 30% MIP; Immediately after 50% MIP; Immediately after 70% MIP
  Assessment of diaphragmatic excursion using ultrasound at 10%, 30%, 50%, and 70% of maximum inspiratory pressure (MIP). Evaluates the diaphragm's mobility as a primary measure of functional response to different inspiratory loads in healthy individuals.

SECONDARY OUTCOMES:
Diaphragmatic thickness at different inspiratory loads | Day 2: Baseline; Immediately after 10% MIP; Immediately after 30% MIP; Immediately after 50% MIP; Immediately after 70% MIP
  Measurement of diaphragmatic thickness using ultrasound at 10%, 30%, 50%, and 70% of maximum inspiratory pressure (MIP). This evaluates muscular response and mobility related to varying inspiratory efforts in healthy subjects.
Diaphragmatic contraction velocity at different inspiratory loads | Day 2: Baseline; Immediately after 10% MIP; Immediately after 30% MIP; Immediately after 50% MIP; Immediately after 70% MIP
  Assessment of diaphragmatic contraction velocity using ultrasound at 10%, 30%, 50%, and 70% of MIP. Evaluates muscular response and mobility during inspiratory efforts.

OTHER OUTCOMES:
Correlation between ultrasound measurements of diaphragmatic function and spirometry parameters | Day 1: Spirometry session, prior to ultrasound evaluations. Day 2: Ultrasound evaluations: Baseline (reposo, pre-load); Immediately after 10% PIM; Immediately after 30% PIM; Immediately after 50% PIM; Immediately after 70% PIM.
  Analysis of the relationship between ultrasound measurements of diaphragmatic function (excursion, thickness, and contraction velocity) and spirometry parameters (such as FEV1, FVC, PEF) obtained in a separate session, to evaluate how ultrasound indicators reflect overall respiratory capacity in healthy individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Eva María Lantarón Caeiro L Dra Eva María Lantarón Caeiro, Dra, Principal Investigator — Universidad de Vigo
Locations (1):
- Facultad de Fisioterapia-Universidade de Vigo, Pontevedra, España, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share IPD has not yet been made. The data will be stored securely and may be considered for sharing in the future, depending on institutional policies, participant consent, and study outcomes.